CLINICAL TRIAL: NCT04977765
Title: Defining the Cardiometabolic Profile of Transgender Boys and Men on Testosterone Therapy
Brief Title: Cardiometabolic Health in Transgender Males
Status: Active, not recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Advancing a Healthier Wisconsin (Unknown)
Responsible Party: Principal Investigator, Susanne Cabrera, Principal Investigator, Medical College of Wisconsin
Other Study IDs: PRO00040486
Record Dates: First submitted 2021-05-25; First posted 2021-07-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Transgender; Transgenderism
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma from participants will be stored and analyzed in labs on the Medical College of Wisconsin campus. All samples will be stored and labeled with coded study identification numbers. Only de-identified samples and data will be shared. The use of these samples will be subject to Medical College of Wisconsin IRB policies and procedures. All specimens and records will be held for a minimum of 10 years from the date of the last entry in the record of the last subject enrolled in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transgender Males: Individuals assigned female gender at birth but considering gender-affirming testosterone therapy. May self-identify as transgender or nonbinary etc.
- Cisgender Controls: Individuals assigned male or female at birth. May identify as cisgender or nonbinary etc. These individuals should not be undergoing or considering any form of hormone therapy.

SUMMARY:
Transgender individuals are those with a gender identity opposite the sex they were assigned at birth. Approximately 1% of the population is transgender, equating to ~60,000 transgender Wisconsinites. A transgender boy or man is someone with a 46,XX karyotype and typical female genitalia but a male gender identity and desire for more male-typical gender expression. Gender-affirming testosterone (hormonal) treatment (GAHT) is the cornerstone of masculinizing therapy for transgender men and boys, resulting in estrogen (E2) suppression and circulating testosterone (T) levels equivalent to cisgender males. Historically, GAHT was initiated after an E2-driven puberty, but the last decade has seen an explosion of referrals for GAHT in transboys, many of whom are exposed to only low E2 levels before puberty is halted with blocker therapy. Knowledge of risks incurred by GAHT rely on low-quality studies, precluding conclusive assessment of GAHT's long-term impact on cardiometabolic outcomes. Data on transboys receiving GAHT before completion of E2-driven puberty are sparser and no studies have addressed mechanisms by which GAHT may affect vascular physiology. The investigators aim to determine the cardiometabolic impact of GAHT in transboys/men and to determine if any differences identified are mechanistically dependent on the timing of GAHT relative to puberty.

DETAILED DESCRIPTION:
Gender-affirming testosterone (hormonal) treatment (GAHT) is the cornerstone of masculinizing therapy for transgender men, resulting in circulating testosterone (T) levels equivalent to cismen and estrogen (E2) suppression. Historically, GAHT was initiated after an E2-driven puberty, but the last decade has seen an explosion of referrals for GAHT in transboys, many of whom are exposed to only low E2 levels before puberty is halted with blocker therapy. Knowledge of risks incurred by GAHT rely on low quality studies, precluding conclusive assessment of GAHT's long-term impact on cardiometabolic outcomes. Data on transboys receiving GAHT before completion of E2-driven puberty are sparser and no studies have addressed mechanisms by which GAHT may affect vascular physiology. The investigators aim to determine the cardiometabolic impact of GAHT in transboys/men and to determine if any differences identified are mechanistically dependent on the timing of GAHT relative to puberty. The vaso-protective benefits of E2 are well-described; higher circulating E2 begins in female puberty, stimulating a long-term increase in the vascular expression of the E2 receptor's alpha isoform (ERα). ERα activation directly stimulates nitric oxide (NO) production from endothelium-derived NO synthase and is critical to maintaining a healthy vascular endothelium. Pre-menopausal women have an increased capacity to produce endothelial NO due to higher E2 levels and vascular ERα expression, resulting in lower cardiovascular disease risk vs age-matched cismen. These data suggest a novel paradigm for the impact of GAHT on vascular health in transmen that differs depending on when GAHT is initiated relative to puberty. The investigators hypothesize that, in transmen who have completed E2-driven puberty, GAHT will induce a regression of vascular endothelial function towards that of cismen by suppressing circulating E2 and ERα expression and that similar regression will not be seen in transboys initiating GAHT prior to pubertal progression. The investigators propose, to our knowledge, a first-of-its-kind longitudinal study of the cardiometabolic impact of 1-year of GAHT in 40 transboys and transmen as compared to cisgender controls with endogenous sex hormones. The impact of GAHT initiation and continuation in transboys/men on in vivo and ex vivo vascular endothelial function, estrogen-stimulated endothelial vasorelaxation, and expression of vascular ERα expression will be determined by measuring changes in conduit vessel endothelium-dependent vasodilation and vascular E2 receptor expression and responsiveness in transboys on puberty blockers and in transmen. The investigators will also determine whether GAHT suppresses the human arteriolar vascular expression of ERα receptors and reduces E2-stimulated endothelial vasorelaxation in transboys/men relative to ciswomen. Secondarily, The investigators will characterize the metabolic, body composition and inflammatory impact of GAHT. This study will provide a novel mechanistic framework for the cardiometabolic impact of GAHT and make available critical information for care providers and patients on how GAHT may affect their cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR TRANSGENDER BOYS AND TRANSGENDER MEN

  1. Sex assigned female at birth and a male gender identity (i.e., transgender male)
  2. Aged 12-30 years
  3. Have a care provider in the Children's Wisconsin Gender Health Clinic or Froedtert Hospital Inclusion Clinic who has determined the individual meets clinical criteria to start testosterone therapy and plans to initiate this therapy
  4. Naïve to testosterone or other masculinizing medical therapy
  5. Cisgender girls/women and transgender boys/men of child-bearing potential (defined as having achieved menarche (first menses), excluding those who have had a hysterectomy or are on GnRH agonist therapy (puberty blockers)) must be willing to use effective birth control (which may include abstinence)) from screening visit until final study visit
  6. Willing and able to give informed consent or have parent or legal guardian provide informed consent if the subject is < 18 years of age

INCLUSION CRITERIA FOR CISGENDER INDIVIDUALS

1. Gender identity concordant with sex assigned at birth (i.e., cisgender)
2. Aged 12-30 years
3. Not related to a transgender participant enrolled in the study
4. Naïve to any sex hormone or pubertal blocker therapy or, specific to cisgender girls/women only, must be ≥ 1 year from use of oral contraceptive or other contraceptive technique (intrauterine device, medroxyprogesterone injections)
5. Willing and able to give informed consent or have parent or legal guardian provide informed consent if the subject is < 18 years of age

INCLUSION CRITERIA FOR OPTIONAL NITROGLYCERIN ENDOTHELIUM-INDEPENDENT VASCULAR FUNCTION STUDY

1. Aged ≥ 18 years
2. No history of migraine headaches
3. Systolic blood pressure ≥ 110 mm Hg
4. No prior past adverse reaction to nitroglycerin
5. Has not used a PDE5 inhibitor (i.e., sildenafil, tadalafil, vardenafil) in the past 7 days

Exclusion Criteria:

-

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Transgender individuals must have been assigned female at birth but identify as transgender/non-binary and interested in gender-affirming testosterone therapy.
Study Population: EXCLUSION CRITERIA FOR TRANSGENDER AND CISGENDER INDIVIDUALS
  1. Any disease affecting glucose, sex steroid, or fat metabolism such as diabetes, polycystic ovary syndrome, or clinical suspicion of insulin resistance)
  2. Any medication use that may affect glucose, sex steroid, or fat metabolism such as metformin or glucocorticoids
  3. Known cardiovascular disease such as hypertension or atherosclerosis
  4. Raynaud's phenomenon or other vascular disease
  5. BMI > 40 kg/m2 for those aged ≥ 18 years or > 95% percentile for age- and sex-assigned at birth in those aged < 18 years
  6. Pregnancy or lactation
  7. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in vascular endothelial function after one year of gender-affirming testosterone therapy as measured by brachial artery ultrasound flow-mediated dilation | 1 year from baseline study visit
  Investigators will examine the effects of gender-affirming testosterone therapy on in vivo endothelial function by brachial artery ultrasound flow-mediated dilation across study visits.
Change in vascular endothelial function after one year of gender-affirming testosterone therapy as measured by by blood pressure. | 1 year from baseline study visit
  Investigators will examine the effects of gender-affirming testosterone therapy on in vivo endothelial function by blood pressure.
Change in vascular endothelial function after one year of gender-affirming testosterone therapy as measured by circulating markers of endothelial activation as measured by plasma analysis | 1 year from baseline study visit
  Investigators will examine the effects of gender-affirming testosterone therapy on in vivo endothelial function by circulating markers of endothelial activation as measured by plasma analysis.

SECONDARY OUTCOMES:
Change in body composition after one year of gender-affirming testosterone therapy as measured by BMI | 1 year from baseline study visit
  Investigators will examine the effect of gender-affirming testosterone therapy on body composition as quantified by body mass index (BMI).
Change in body composition after one year of gender-affirming testosterone therapy as measured by DXA scans. | 1 year from baseline study visit
  Investigators will examine the effect of gender-affirming testosterone therapy on body composition as quantified by total body dual-energy X-ray absorptiometry (DXA) scan which provides information about the amount and distribution of fat and muscle in the body.
Change in body composition after one year of gender-affirming testosterone therapy as measured by the ratio of waist-to-hip circumference. | 1 year from baseline study visit
  Investigators will examine the effect of gender-affirming testosterone therapy on body composition as quantified by the ratio of waist-to-hip circumference which provides information about the amount and distribution of fat and muscle in the body.
Change in lipid profile after one year of gender-affirming testosterone therapy | 1 year from baseline study visit
  Investigators will measure the effect of gender-affirming testosterone therapy on the various components of a fasting lipid profile (triglyceride level, HDL, LDL, and total cholesterol).
Change in systemic inflammation after one year of gender-affirming testosterone therapy | 1 year from baseline study visit
  Investigators will examine the effect of gender-affirming testosterone therapy on circulating levels of inflammatory cytokines as measured by plasma analysis.
Change in glucose metabolism after one year of gender-affirming testosterone therapy as measured by fasting insulin level in the blood. | 1 year from baseline study visit
  Investigators will examine the effect of gender-affirming testosterone therapy on fasting insulin.
Change in glucose metabolism after one year of gender-affirming testosterone therapy as measured by fasting blood glucose level. | 1 year from baseline study visit
  Investigators will examine the effect of gender-affirming testosterone therapy on fasting glucose.
Change in glucose metabolism after one year of gender-affirming testosterone therapy as measured by HbA1c | 1 year from baseline study visit
  Investigators will examine the effect of gender-affirming testosterone therapy on HbA1c levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States